CLINICAL TRIAL: NCT07379151
Title: Evaluation of the Antibody Persistence in African Participants Beyond Five Years After Immunization With MenFiveTM (NmCV-5), a Pentavalent Meningococcal ACYWX Conjugate Vaccine
Brief Title: Evaluation of the Antibody Persistence Beyond Five Years After Immunization With MenFiveTM (NmCV-5), a Pentavalent Meningococcal ACYWX Conjugate Vaccine
Acronym: PERS-ACYWX-03
Status: Not yet recruiting | Type: Observational
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: PERS-ACYWX-03
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Meningoccocal Disease
Keywords: Seropersistence; Meningococcal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NmCV-5
- MenACWY-D

SUMMARY:
This study will measure immune persistence of the NmCV-5 more than 5 years after a single dose vaccination in participants 2-29 years of age in Mali and The Gambia.

DETAILED DESCRIPTION:
This non-interventional long-term follow-up study will involve one telephonic contact in all 1800 former participants from study ACYWX-03 followed by one visit beyond five years after vaccination in a subset of 450 participants. This subset will be randomly selected to participate in a follow-on immune persistence evaluation. To document the duration of the immune response and any requirement of booster dose in the target population, this study is intended to explore antibody persistence.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and assent (if applicable)

Exclusion Criteria:

* Current or previous, confirmed disease caused by Neisseria meningitidis at any given time since meningococcal vaccination
* Any condition or criteria that in the opinion of the investigator might compromise the well-being of the participant or the compliance with study procedures or interfere with the outcome of the study

Ages: 7 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants from the previous study ACYWX-03 conducted at the Gambia and Mali
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titers (GMTs) measured by rSBA against serogroups A, C, Y, W and X | five-six years after vaccination.

SECONDARY OUTCOMES:
Percentage of participants with rSBA titers ≥ 8 | five-six years after vaccination.
Percentage of participants with rSBA titers ≥ 128 | five-six years after vaccination

IPD SHARING:
Plan to Share IPD: No